CLINICAL TRIAL: NCT01342146
Title: Efficiency and Safety of Pegylated Somatropin(PEG-somatropin) in the Treatment of Children With Growth Hormone Deficiency: a Multicenter, Randomized, Open-label, Controlled Phase 2 Study
Brief Title: Efficiency and Safety Study of Pegylated Somatropin to Treat Growth Hormone Deficiency Children
Acronym: PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Huazhong University of Science and Technology (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Capital Medical University (Other); Children's Hospital of Fudan University (Other)
Responsible Party: International Regulatory Affairs Department, GeneScience Pharmaceuticals Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci-004 CT
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2011-05

CONDITIONS: Growth Hormone Deficiency
Keywords: pegylated Somatropin; PEG-GH; Growth hormone; PEG-rhGH; Growth hormone deficiency (GHD); Phase 2 study
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pegylated Somatropin — 0.1 mg/kg/wk once a week for 25 weeks
  Other Names: PEG-rhGH,PEG-growth hormone,PEG-Somatropin
Drug: pegylated Somatropin — 0.2 mg/kg/wk once a week for 25 weeks
  Other Names: PEG-rhGH,PEG-growth hormone,PEG-Somatropin
Drug: Jintropin AQ — 0.25 mg/kg/wk, once a day for 25 weeks
  Other Names: Somatropin injectable solution,rhGH injection

SUMMARY:
The purpose of the multicenter, randomized, open-label, controlled phase II study is to determine whether pegylated recombinant human growth hormone is effective in the treatment of children with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* have a height less than two standard deviations (SD) below the median height for individuals of the same age or height, a growth velocity (GV) ≤4 cm/yr, a GH peak concentration <7 ng/ml in two different provocative tests, a bone age (BA; ≤9 years in girls and ≤10 years in boys) at least 2 years less than his/her chronological age (CA);
* be in preadolescence (Tanner stage 1) and have a CA >3 years;
* have a height value recorded 3 months before the start of GH treatment to calculate pre-treatment GV;
* receive no prior GH treatment.
* sign informed consent

Exclusion Criteria:

* patients with severe cardiopulmonary
* patients with hematological diseases
* a current or past history of malignant tumors
* immunodeficiency diseases
* mental diseases
* patients positive for hepatitis B e-antibody (HBeAb)
* hepatitis B surface antigen (HBsAg)
* hepatitis B e antigen (HBeAg)
* patients with other growth disorders, such as Turner syndrome
* constitutional delay of growth and puberty, and Laron syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Growth velocity | 25 weeks

SECONDARY OUTCOMES:
height standard deviation score for chronological age (Ht SDSCA) | 25 weeks
IGF-1 | 25 weeks
IGFBP3 | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, Doctor, Principal Investigator — Tongji Hospital

REFERENCES:
- [Result] Luo X, Hou L, Liang L, Dong G, Shen S, Zhao Z, Gong CX, Li Y, Du ML, Su Z, Du H, Yan C. Long-acting PEGylated recombinant human growth hormone (Jintrolong) for children with growth hormone deficiency: phase II and phase III multicenter, randomized studies. Eur J Endocrinol. 2017 Aug;177(2):195-205. doi: 10.1530/EJE-16-0905. Epub 2017 May 31. PMID 28566441